CLINICAL TRIAL: NCT05182099
Title: AIRTM Deep Learning Reconstruction of Abdominal High Resolution Gd-EOB-DTPA Enhanced MRI in Patients With Suspicious Focal Liver Lesions: Image Quality Assessment
Brief Title: High Resolution HBA-MRI Using Deep Learning Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2021-3044
Record Dates: First submitted 2021-12-16; First posted 2022-01-10 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Liver Diseases; Magnetic Resonance Imaging; Deep Learning
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: blinded to the reconstruction types
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional image reconstruction (Other): Gd-EOB-DTPA enhanced liver MRI images are reconstructed using a conventional image reconstruction algorithm. It is automatically generated from a MRI console after the examination.
  Interventions: Diagnostic Test: Liver MRI
- Deep learning image reconstruction (Active Comparator): Gd-EOB-DTPA enhanced liver MRI images are reconstructed using a deep learning based image reconstruction algorithm (AIRTM). It is additionally generated aside from the conventional images.
  For obtaining the images, we will use the same MRI raw data which is used for conventional image reconstruction.
  Interventions: Diagnostic Test: Liver MRI

INTERVENTIONS:
Diagnostic Test: Liver MRI — Gd-EOB-DTPA enhanced MRI consists of T2-weighted image (T2WI), diffusion weighted image (DWI) and precontrast T1-weighted image (T1WI), dynamic T1WI (arterial, portal and transitional phases), and hepatobiliary phase.

SUMMARY:
This study aims to compare image qualities between conventionally reconstructed MRI sequences and deep-learning reconstructed MRI sequences from the same data in patients who undergo Gd-EOB-DTPA enhanced liver MRI. The AIRTM deep learning sequence is applicable for various MRI sequences including T2-weighted image (T2WI), T1-weighted image and diffusion-weighted image (DWI). We plan to perform intra-individual comparisons of the image qualities between two reconstructed image datasets.

ELIGIBILITY:
Inclusion Criteria:

* older than 20 years old
* scheduled for Gd-EOB-DTPA enhanced liver MRI at a 3T scanner (Premier, GE Healthcare) in our institution
* signed informed consent

Exclusion Criteria:

* younger than 20 years old
* any absolute/relative contrast indication of Gd-EOB-DTPA enhanced MRI
* history of transient dyspnea after Gd-EOB-DTPA administration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall image quality of arterial phase | 3 months after enrollment completion
  qualitative assessment of arterial phase on a five point scale (highest score indicates better image quality)

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No